CLINICAL TRIAL: NCT00021814
Title: Medical Therapy of Prostatic Symptoms
Acronym: MTOPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTOPS (completed); U01DK046472 (NIH)
Record Dates: First submitted 2001-08-04; First posted 2001-08-06 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Prostatic Hyperplasia; Prostatic Hypertrophy, Benign
Keywords: BPH progression; Medical Therapy; Finasteride; Doxazosin; Randomized; Multi-center; Clinical Trial; Proscar; Cardura
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Doxazosin; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Doxazosin and Finasteride placebos
  Interventions: Drug: Doxazosin placebo; Drug: Finasteride placebo
- Doxazosin (Experimental): Doxazosin and Finasteride placebo
  Interventions: Drug: Doxazosin; Drug: Finasteride placebo
- Finasteride (Experimental): Doxazosin placebo and Finasteride
  Interventions: Drug: Finasteride; Drug: Doxazosin placebo
- Combination (Experimental): Doxazosin and Finasteride
  Interventions: Drug: Doxazosin; Drug: Doxazosin placebo

INTERVENTIONS:
Drug: Doxazosin
  Arms: Combination; Doxazosin
Drug: Finasteride
  Arms: Finasteride
Drug: Doxazosin placebo
  Arms: Combination; Finasteride; Placebo
Drug: Finasteride placebo
  Arms: Doxazosin; Placebo

SUMMARY:
The Medical Therapy of Prostatic Symptoms (MTOPS) is a clinical research study sponsored by the National Institutes of Health (NIH). The study will test whether the oral drugs finasteride (Proscar) and doxazosin (Cardura), alone or together, can delay or prevent further worsening of symptoms in men with Benign Prostatic Hyperplasia (BPH).

MTOPS is the largest and longest study to simultaneously test whether these drugs can delay or prevent the clinical progression (symptom worsening) of BPH. Seventeen U.S. medical centers recruited 2,931 men diagnosed with symptomatic BPH between December 1995 and March 1998. Study doctors will continue to follow these men through November 2001 on a quarterly basis. In addition to the clinical progression of BPH, MTOPS will include evaluations of prostate volume by ultrasound, prostate biopsies among a subgroup of volunteers, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Peak urinary flow rate at least 4 ml/sec but not greater than 15 ml/sec; and voided volume is at least 125 ml.
* American Urological Association Symptom Score is greater than or equal to 8 and less than or equal to 30.
* Voluntarily signed the informed consent agreement prior to the performance of any study procedures.

Exclusion Criteria:

* Serum prostate specific antigen level greater than 10 ng/ml.
* Supine blood pressure less than 90/70 mmHG. Orthostatic hypotension.
* Any prior medical or surgical intervention for BPH.
* Received any prior experimental intervention (either medical or surgical) for prostate disease or enrolled in any other study protocol.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3407 (Actual)
Dates: Start 1995-12 (Actual); Primary Completion 2001-11-30 (Actual); Study Completion 2001-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. David Crawford, Principal Investigator — Clinic 01 - Univ of Colorado Health Sciences Center; Steven A. Kaplan, Principal Investigator — Clinic 02 - New York Presbyterian Hospital; Claus Roehrborn, Principal Investigator — Clinic 03 - UT Southwestern Medical Center; Noah S. Schenkman, Principal Investigator — Clinic 04 - Walter Reed Army Medical Center; Herbert Lepor, Principal Investigator — Clinic 06 - New York University School of Medicine; Kevin M. Slawin, Principal Investigator — Clinic 07 - Baylor College of Medicine; John P. Foley, Principal Investigator — Clinic 08 - Brooke Army Medical Center; Joe W. Ramsdell, Principal Investigator — Clinic 09 - University of California San Diego; Mani Menon, Principal Investigator — Clinic 10 - Henry Ford Hospital; Michael M. Lieber, Principal Investigator — Clinic 11 - Mayo Foundation; Kevin T. McVary, Principal Investigator — Clinic 12 - Northwestern University; Joseph A. Smith, Principal Investigator — Clinic 13 - Vanderbilt University; Gerald L. Andriole, Principal Investigator — Clinic 14 - Washington University; Harris E. Foster, Principal Investigator — Clinic 15 - Yale University; Harry S. Clarke, Principal Investigator — Clinic 16 - Emory University; Karl J. Kreder, Principal Investigator — Clinic 17 - University of Iowa; Stephen C. Jacobs, Principal Investigator — Clinic 18 - University of Maryland; Gary J. Miller, Principal Investigator — Diagnostic Center - Univ of Colorado Health Sciences Center; Oliver M. Bautista, Principal Investigator — Biostatistical Coordinating Center - George Washington Univ.
Locations (17):
- United States (17):
  - University of California, La Jolla, California
  - Univ of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Health Systems, Detroit, Michigan
  - Mayo Foundation, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data and specimens will be submitted to the NIDDK Central Repository
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2006
URL: https://repository.niddk.nih.gov/studies/mtops/?query=mtops

REFERENCES:
- [Background] Berry SJ, Coffey DS, Walsh PC, Ewing LL. The development of human benign prostatic hyperplasia with age. J Urol. 1984 Sep;132(3):474-9. doi: 10.1016/s0022-5347(17)49698-4. PMID 6206240
- [Background] Sidney S, Quesenberry CP Jr, Sadler MC, Guess HA, Lydick EG, Cattolica EV. Incidence of surgically treated benign prostatic hypertrophy and of prostate cancer among blacks and whites in a prepaid health care plan. Am J Epidemiol. 1991 Oct 15;134(8):825-9. doi: 10.1093/oxfordjournals.aje.a116157. PMID 1719806
- [Background] Gormley GJ, Stoner E, Bruskewitz RC, Imperato-McGinley J, Walsh PC, McConnell JD, Andriole GL, Geller J, Bracken BR, Tenover JS, et al. The effect of finasteride in men with benign prostatic hyperplasia. The Finasteride Study Group. N Engl J Med. 1992 Oct 22;327(17):1185-91. doi: 10.1056/NEJM199210223271701. PMID 1383816
- [Background] Lepor H, Gup DI, Baumann M, Shapiro E. Laboratory assessment of terazosin and alpha-1 blockade in prostatic hyperplasia. Urology. 1988 Dec;32(6 Suppl):21-6. PMID 2462301
- [Background] Lepor H, Henry D, Laddu AR. The efficacy and safety of terazosin for the treatment of symptomatic BPH. Prostate. 1991;18(4):345-55. doi: 10.1002/pros.2990180408. PMID 1711689
- [Background] Guess HA. Benign prostatic hyperplasia: antecedents and natural history. Epidemiol Rev. 1992;14:131-53. doi: 10.1093/oxfordjournals.epirev.a036083. No abstract available. PMID 1283852
- [Background] McConnell JD. Androgen ablation and blockade in the treatment of benign prostatic hyperplasia. Urol Clin North Am. 1990 Aug;17(3):661-70. PMID 1695786
- [Background] Barry MJ. Epidemiology and natural history of benign prostatic hyperplasia. Urol Clin North Am. 1990 Aug;17(3):495-507. PMID 1695778
- [Background] Mebust WK, Holtgrewe HL, Cockett AT, Peters PC. Transurethral prostatectomy: immediate and postoperative complications. A cooperative study of 13 participating institutions evaluating 3,885 patients. J Urol. 1989 Feb;141(2):243-7. doi: 10.1016/s0022-5347(17)40731-2. PMID 2643719
- [Result] McConnell JD, Roehrborn CG, Bautista OM, Andriole GL Jr, Dixon CM, Kusek JW, Lepor H, McVary KT, Nyberg LM Jr, Clarke HS, Crawford ED, Diokno A, Foley JP, Foster HE, Jacobs SC, Kaplan SA, Kreder KJ, Lieber MM, Lucia MS, Miller GJ, Menon M, Milam DF, Ramsdell JW, Schenkman NS, Slawin KM, Smith JA; Medical Therapy of Prostatic Symptoms (MTOPS) Research Group. The long-term effect of doxazosin, finasteride, and combination therapy on the clinical progression of benign prostatic hyperplasia. N Engl J Med. 2003 Dec 18;349(25):2387-98. doi: 10.1056/NEJMoa030656. PMID 14681504
- [Result] Kusek JW, Ahrens A, Burrows PK, Clarke HS, Foster HE, Hanson K, Jacobs SC, Kirkemo A, O'Berry K, Pavlik VN; MTOPS Research Group. Recruitment for a clinical trial of drug treatment for benign prostatic hyperplasia. Urology. 2002 Jan;59(1):63-7. doi: 10.1016/s0090-4295(01)01454-6. PMID 11796283
- [Result] Bautista OM, Kusek JW, Nyberg LM, McConnell JD, Bain RP, Miller G, Crawford ED, Kaplan SA, Sihelnik SA, Brawer MK, Lepor H. Study design of the Medical Therapy of Prostatic Symptoms (MTOPS) trial. Control Clin Trials. 2003 Apr;24(2):224-43. doi: 10.1016/s0197-2456(02)00263-5. PMID 12689743
- [Derived] Long B, Cheema A, Copelan O, Joyce C, Feffer M, McVary KT. Five-Year Outcomes of Water Vapor Therapy vs Doxazosin, Finasteride, and Combination Therapy for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: Cohort Data From the Medical Therapy of Prostatic Symptoms Trial. Urology. 2025 Dec;206:142-149. doi: 10.1016/j.urology.2025.07.016. Epub 2025 Jul 17. PMID 40683564
- See also: MTOPS public access site. Userid and password not required. — http://www.bsc.gwu.edu/mtops/index.html